CLINICAL TRIAL: NCT00497315
Title: A Randomized Multicenter Phase II Study Of Induction Therapy With Pemetrexed And Cisplatin Followed By Chemoradiation With Pemetrexed Versus Chemoradiation With Pemetrexed Followed By Consolidation Therapy With Pemetrexed And Cisplatin In Patients With Stage III Non-Small Cell Lung Cancer: Paccora Trial
Brief Title: Evaluation of Pemetrexed Combined With Cisplatin and Radiotherapy for Unresectable Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: PACCORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Eli Lilly and Company (Industry)
Responsible Party: Thoracic Oncology Group Antwerp - Paul Germonpre, Thoracic Oncology Group Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOGA 0502; Eudra CT 2005-004030-40
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Chemoradiation; locally advanced NSCLC; pemetrexed; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Drug Therapy, Combination; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): pemetrexed + cisplatin (3 cycles) followed by thoracic irradiation + pemetrexed
  Interventions: Drug: combination chemotherapy (pemetrexed + cisplatin); Radiation: thoracic irradiation + pemetrexed
- B (Experimental): thoracic irradiation + pemetrexed followed by pemetrexed + cisplatin
  Interventions: Drug: combination chemotherapy (pemetrexed + cisplatin); Radiation: thoracic irradiation + pemetrexed

INTERVENTIONS:
Drug: combination chemotherapy (pemetrexed + cisplatin) — pemetrexed 500 mg/m2 + cisplatin 75 mg/m2 (q 3 weeks for 3 cycles)
  Other Names: Alimta
Radiation: thoracic irradiation + pemetrexed — pemetrexed 500 mg/m2 (q 3weeks for 2 cycles), 60 GY (30 fractions of 2 GY)
  Other Names: Alimta

SUMMARY:
The aim of this study is to evaluate if the multi modality treatment pemetrexed combined with cisplatin and radiotherapy can lead to a better tumor control and/or a better side-effect profile in patients with locally advanced NSCLC. Patients will be randomized between 3 cycles of induction chemotherapy followed by concurrent chemoradiotherapy or concurrent chemoradiotherapy followed by 3 cycles of adjuvant combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* cytological or histological proven NSCLC
* unresectable stage III NSCLC
* presence of at least one measurable lesion (RECIST criteria)
* adequate haematological, renal and hepatic function
* adequate lung function reserve
* good condition, weight loss <10 % over previous 6 months, life expectancy > 3 months

Exclusion Criteria:

* previous chemo- or radiotherapy for NSCLC
* distant metastasis or a malignant pleural or pericardial effusion
* second active primary malignancy or serious concomitant medical disease
* interstitial lung disease
* auto-immune systemic disease with potential involvement of the lungs
* inability to interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5-day period
* concomitant use of amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Response rate | after each treatment modality and 5 year follow-up

SECONDARY OUTCOMES:
Toxicity | at the end of each cycle and 5 year follow-up
Time to progression | 5 year follow-up
Overall survival | median survival and 2-year survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Germonpre, MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - ZNA Middelheim, Antwerp, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp
  - St Augustinus Ziekenhuis, Wilrijk, Antwerp